CLINICAL TRIAL: NCT06985199
Title: AHOMKA Qualitative Study For Adaptation of the Medtronic Empower Health Platform
Brief Title: Culturally-adapted Mobile Health Intervention for Hypertension Care
Acronym: AHOMKA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: University of Ghana Medical School (Other); Beth Israel Deaconess Medical Center (Other); University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00001929
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
Keywords: hypertension, mobile health
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Feasibility study of mobile health application
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced Usual Care Group (Experimental): Participants with uncontrolled hypertension and the owner of a cell phone are selected. Participants will receive usual care as determined by their provider.
  Interventions: Behavioral: Enhanced Usual Care Group

INTERVENTIONS:
Behavioral: Enhanced Usual Care Group — A culturally-adapted mobile health platform will be used in the intervention to enable participants to record blood pressure and heart rate readings at home and store data in the mobile platform. Providers will have access to the store data using a provider-facing app.

SUMMARY:
A single-arm study to assess the ability of the AHOMKA platform for hypertension management to affect blood pressure change among urban and rural patients in Ghana.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hypertension

Exclusion Criteria:

* Comorbidities

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure levels from Baseline | Baseline, 6 months
  Changes in blood pressure levels, measured in mmHg, will be assessed at the baseline and 6-month endline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Valencia Koomson, Principal Investigator — Tufts University; Mark Tettey, MD, Principal Investigator — University of Ghana
Locations (2):
- Ghana (2):
  - National Cardiothoracic Center, Accra, Ghana
  - Cardiothoracic Center - Outpatient Department, Ho, Ghana

IPD SHARING:
Plan to Share IPD: No